CLINICAL TRIAL: NCT04277442
Title: A Pilot Study of Nivolumab in Combination With Decitabine and Venetoclax in TP53-Mutated Acute Myeloid Leukemia
Brief Title: Testing Nivolumab in Combination With Decitabine and Venetoclax in Patients With Newly Diagnosed TP53 Gene Mutated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-01125; NCI-2020-01125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU 19305; 10317 (Other: Ohio State University Comprehensive Cancer Center LAO); 10317 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Results first posted 2024-10-22 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine; Injections; Nivolumab; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab, decitabine, venetoclax) (Experimental): INDUCTION: Patients receive nivolumab IV over 30 minutes on day 15 of cycle 1 and days 1 and 15 of subsequent cycles, decitabine IV over 60 minutes on days 1-10 of induction cycle 1 (and cycles 2 and 3 if needed), and venetoclax PO QD on days 1-21. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients who achieve a CR or CRi receive nivolumab IV over 30 minutes on days 1 and 15, decitabine IV over 60 minutes on days 1-5, and venetoclax PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Biological: Nivolumab; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
Drug: Venetoclax — Given PO
  Other Names: ABT 199; ABT-0199; ABT-199; ABT199; GDC 0199; GDC-0199; GDC0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This trial studies the side effects of nivolumab in combination with decitabine and venetoclax and to see how well they work in treating patients with TP53-mutated acute myeloid leukemia. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as decitabine and venetoclax, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. This study is being done to find out whether giving nivolumab, decitabine, and venetoclax is better or worse than the usual approach for TP53-mutated acute myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary data regarding the safety and tolerability of decitabine and venetoclax in combination with nivolumab when given for frontline therapy in TP53 mutated acute myeloid leukemia (AML) patients.

II. To obtain preliminary data regarding the rate of complete remission (CR), complete remission with incomplete hematological recovery (CRh), and complete remission with incomplete count recovery (CRi) in TP53 mutated AML who are treated with decitabine and venetoclax in combination with nivolumab for frontline therapy.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To obtain preliminary data regarding progression free survival (PFS) for TP53 mutated AML patients receiving combination therapy.

III. To obtain preliminary data regarding the overall survival (OS) for TP53 mutated patients receiving this combination therapy.

IV. To obtain preliminary data regarding minimal residual disease through monitoring TP53 mutational burden prior and throughout treatment.

V. To obtain preliminary data regarding the frequency of graft versus host disease (GVHD) including veno-occlusive disease (VOD) in patients who subsequently receive allogeneic transplantation after this combination therapy.

OUTLINE:

INDUCTION: Patients receive nivolumab intravenously (IV) over 30 minutes on day 15 of cycle 1 and days 1 and 15 of subsequent cycles, decitabine IV over 60 minutes on days 1-10 of induction cycle 1 (and cycles 2 and 3 if needed), and venetoclax orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients who achieve a CR or CRi receive nivolumab IV over 30 minutes on days 1 and 15, decitabine IV over 60 minutes on days 1-5, and venetoclax PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed acute myeloid leukemia (AML)
* Presence of TP53 mutation at diagnosis
* Newly diagnosed, untreated AML
* Patients who received prior hypomethylating therapy for a prior myelodysplastic syndrome (MDS) diagnosis are allowed
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN), (except for patients with Gilbert's disease)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 x institutional ULN
* Glomerular filtration rate (GFR) > 40 mL/min/1.73 m^2
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better. A baseline troponin should be within normal limits and baseline oxygen saturation should be greater than or equal to 92%. A baseline electrocardiogram (ECG) should be normal, or with stable changes if patient has chronic ECG changes
* Active infection is permitted if the infection is under control
* White blood count (WBC) must be =< 25,000 at time of day 1 of study treatment. Cytoreduction with Hydrea and leukapheresis is allowed
* Risks from venetoclax and nivolumab to the developing human fetus cannot be ruled out. For this reason and because decitabine is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Contraception use should be continued 6 months after the completion of all study treatments for women of child bearing potential. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 7 months after completion of decitabine, venetoclax, or nivolumab administration
* Ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making are allowed to participate as long as the patient has a legally authorized representative (LAR) or caregiver

Exclusion Criteria:

* Patients with history of prior allogeneic transplantation. This is due to this being a pilot study with a limited number of patients
* Patients with known autoimmune disease. Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption). Physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients with hyperleukocytosis requiring immediate cytoreductive chemotherapy (WBC >= 100,000 with symptoms of leukostasis)
* Isolated extramedullary leukemia of central nervous system (CNS) involvement with leukemia
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to decitabine, venetoclax, or nivolumab
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because fetal risk has been demonstrated with decitabine with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with decitabine, breastfeeding should be discontinued if the mother is treated with decitabine. These potential risks may also apply to other agents used in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-05-12 (Actual); Study Completion 2022-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice S Mims, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nivolumab, Decitabine, Venetoclax): INDUCTION: Patients receive nivolumab IV over 30 minutes on day 15 of cycle 1 and days 1 and 15 of subsequent cycles, decitabine IV over 60 minutes on days 1-10 of induction cycle 1 (and cycles 2 and 3 if needed), and venetoclax PO QD on days 1-21. Treatment repeats every 28 days for up to 3 cycles in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE: Patients who achieve a CR or CRi receive nivolumab IV over 30 minutes on days 1 and 15, decitabine IV over 60 minutes on days 1-5, and venetoclax PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Decitabine: Given IV
  Nivolumab: Given IV
  Venetoclax: Given PO
Period: Overall Study
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Started | 1
Completed | 0
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Toxicity will be graded and reported according to the revised National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.
Time Frame: Up to day 15 of cycle 1 (each cycle is 28 days)
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
participants
  Neutropenic Fever | 1
  Fatigue | 1
  Edema face | 1
  Diarrhea | 1
  Mucositis oral | 1
  Dyspnea | 1
  Cough | 1
  Electrocardiogram QT corrected interval prolonged | 1
  Hematuria | 1
  Proteinuria | 1
  Hyponatremia | 1
  Blood bilirubin increased | 1
  Alkaline phosphatase increased | 1
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Blood lactate dehydrogenase increased | 1
  INR increased | 1
  Anemia | 1
  Urinary tract infection | 1
  Febrile neutropenia | 1
  Confusion | 1
  Bacteremia | 1
  Epistaxis | 1
  Nausea | 1
  Vomiting | 1
  Hypophosphatemia | 1
  Hypoalbuminemia | 1
  Activate partial thromboplastin time prolonged | 1
  White blood cell decreased | 1
  Platelet count decreased | 1
  Neutrophil count decreased | 1
  Lymphocyte count decreased | 1
  Hypocalcemia | 1
  Thromboembolic event | 1
  Chills | 1
  Lung infection | 1
  Hypothermia | 1
  Thrush | 1
  Anorexia | 1

2. Primary Outcome: Number of Patients That Are Able to Complete 3 Cycles of Therapy
Description: Feasibility will be met if 10 of 13 patients are able to complete 3 cycles of therapy.
Time Frame: Up to day 15 of cycle 1 (each cycle is 28 days)
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
participants | 0

3. Primary Outcome: Response
Description: Response will be defined as being able to achieve complete remission, complete remission with incomplete count recovery, or complete remission with incomplete hematological recovery by cycle 3.
Time Frame: Up to day 15 of cycle 1 (each cycle is 28 days)
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
participants | 0

4. Secondary Outcome: Anti-tumor Activity
Description: Patients will be carefully monitored for tumor response and symptom relief in addition to safety and tolerability. Data that are collected serially over time will be explored graphically using box plots and/or individual time plots as well as analytically with either repeated measures analysis of variance or Friedman's nonparametric test.
Time Frame: Up to 3 years
Population: Data was not collected due to low enrollment
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 0

5. Secondary Outcome: Progression-free Survival
Description: 95% confidence intervals will be given.
Time Frame: Up to 2 years 5 months
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
participants | 0

6. Secondary Outcome: Overall Survival
Description: 95% confidence intervals will be given.
Time Frame: Up to 2 years 5 months
Measure: Number; unit: participants
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 1
participants | 0

7. Secondary Outcome: Minimal Residual Disease (MRD)
Description: Will assess MRD by measuring the TP53 mutational burden with variant allele frequency before and after response is achieved to see if there is a change. Will also evaluate its association with MRD status at each time point using chi-square test of independence.
Time Frame: Up to 3 years
Population: Data not collected due to low enrollment
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 0

8. Secondary Outcome: T Cell Response
Description: Will study the T cell response against both tumor associated antigen and tumor specific antigen. Analyses of the data will be primarily descriptive in nature given the relatively small sample size.
Time Frame: Up to 3 years
Population: Data not collected and analyzed due to low enrollment
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 0

9. Secondary Outcome: Deoxyribonucleic Acid (DNA) Methylation
Description: Will study the level of global DNA methylation as well as methylation levels of specific genes involved in immune checkpoint, such as PD-L1, PD-L2, PD-1 and CTLA4. Analyses of the data will be primarily descriptive in nature given the relatively small sample size.
Time Frame: Up to 3 years
Population: Data not collected or analyzed due to low enrollment
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Patients were evaluated for Adverse Events from the start of study to study completion using the NCI CTCAE version 5.0 for up to 2 years 5 months.
Arm/Group | Treatment (Nivolumab, Decitabine, Venetoclax)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Decitabine, Venetoclax) (N=1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nivolumab, Decitabine, Venetoclax) (N=1)
Fatigue (General disorders) | 1 (1)
Edema Face (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Electrocardiogram QT corrected Interval prolonged (Investigations) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Blood bilirubin Increased (Investigations) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Blood lactate dehydrogena se Increased (Investigations) | 1 (1)
NR Increased (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Thromboembolic (Vascular disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-08-16): https://cdn.clinicaltrials.gov/large-docs/42/NCT04277442/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT04277442/ICF_001.pdf